CLINICAL TRIAL: NCT04140812
Title: STRATifying Risk for intracErebral haemorrhaGe and Neurodevelopmental DIsorders in Newborns
Brief Title: Stratifying Risk for Intracerebral Haemorrhage
Acronym: NEW_STRATEGI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 294_19B
Record Dates: First submitted 2019-10-21; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Preterm Birth; Coagulation Protein Disorders; Coagulation Disorder Neonatal
Keywords: Preterm; Coagulation; LC-MS/MS; ICH; IVH; Neonatal
MeSH Terms: conditions — Premature Birth; Coagulation Protein Disorders; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Term infants (≥37+0 weeks) (Active Comparator): Blood collection (5 drops) during newborn-screening (36-72h after birth) or postnatal hospitalization (<36h after birth). The blood sample will then be examined using mass spectrometry (LC-MS/MS).
  Interventions: Diagnostic Test: mass spectrometry (LC-MS/MS)
- Preterm infants (≤32+0 weeks) (Experimental): Blood collection (5 drops) during newborn-screening (36-72h after birth) or postnatal hospitalization (<36h after birth). The blood sample will then be examined using mass spectrometry (LC-MS/MS).
  Interventions: Diagnostic Test: mass spectrometry (LC-MS/MS)

INTERVENTIONS:
Diagnostic Test: mass spectrometry (LC-MS/MS) — Blood collection (5 drops) during newborn-screening (36-72h after birth) or postnatal hospitalization (<36h after birth). The blood sample will then be examined using mass spectrometry (LC-MS/MS) for 125 proteins.

SUMMARY:
This study aims to investigates the role of gestational age on the prevalence of coagulation factors and components of the complement system in preterm- (≤32+0 weeks) and term neonates (≥37+0 weeks) and their role for the development of brain hemorrhage.

DETAILED DESCRIPTION:
The occurrence of brain hemorrhage (germinal matrix hemorrhage and intraventricular hemorrhage, GM-IVH) in newborns, especially in preterm infants, is one of the most important prognostic factors for mortality and morbidity (especially for later neurological development) in this collective. The risk of high-grade bleeding in extremely premature infants (22 weeks) is approx. 38% and decreases to approx. 7% by the 28th week. The total frequency of GM-IVH is around 8% in gestational weeks 23 to 31, with each additional gestational week reducing the risk by 3.5%. The etiopathology of brain hemorrhage is complex and involves both environmental and genetic factors. Recent studies particularly suggest an involvement of the immature coagulation system in preterm neonates. Global coagulation parameters, such as the International Normalized Ratio (INR), have already been associated with an increased risk of bleeding, but rarely show fluctuations outside the norm. Furthermore, polymorphisms in the area of individual coagulation factors as well as other inflammatory and vascular individual components of coagulation, are associated with an increased risk of bleeding. Mass spectrometry has long been used for the analysis of biological samples and has developed into an indispensable tool for proteomics research. The study aims to establish the mass spectrometric detection of a total of 125 blood plasma factors containing the individual components of the coagulation system and the complement system. The method enables quantitative detection of the coagulation system with even the smallest sample quantities, so that sampling can be combined with routine measures, particularly in the field of neonatology. This pilot study to compare the compositional differences regarding coagulation factors and the complement system in relation to the gestational age (i.e. preterm ≤32+0 weeks vs. term neonates ≥37+0 weeks).

ELIGIBILITY:
Inclusion Criteria:

* medical indication (newborn screening) and informed consent for blood drawing

Exclusion Criteria:

* clinical evidence of infection
* clinical evidence of hyperbilirubinemia
* Preeclampsia (PE), HELLP-syndrome, intrauterine growth restriction (IUGR) and PE+IUGR

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite mass spectrometric profile of coagulation and complement factors stratified by preterm/term neonates. | Single time point (1 day)
  Individual composite mass spectrometric profile of 125 blood plasma factors containing the individual components of the coagulation system and the complement system of term (≥37+0 SSW) compared to preterm neonates (≤32+0 SSW)

OTHER OUTCOMES:
Composite mass spectrometric profile of coagulation and complement factors stratified by gestational week | Single time point (1 day)
  Individual composite mass spectrometric profile of 125 blood plasma factors containing the individual components of the coagulation system and the complement system stratified by gestational week
Composite mass spectrometric profile of coagulation and complement factors stratified by gender | Single time point (1 day)
  Individual composite mass spectrometric profile of 125 blood plasma factors containing the individual components of the coagulation system and the complement system of female compared to male neonates
Composite mass spectrometric profile of coagulation and complement factors correlated to body weight | Single time point (1 day)
  Individual composite mass spectrometric profile of 125 blood plasma factors containing the individual components of the coagulation system and the complement system correlated to body weight
Composite mass spectrometric profile of coagulation and complement factors stratified by medication | Single time point (1 day)
  Individual composite mass spectrometric profile of 125 blood plasma factors containing the individual components of the coagulation system and the complement system stratified by perinatal medication to non-perinatal medication.
Mass spectrometric profile of coagulation and complement factors correlated to CRP | Single time point (1 day)
  Individual mass spectrometric profile of 125 blood plasma factors containing the individual components of the coagulation system and the complement system correlated to C-reaktive Protein (CRP)
Mass spectrometric profile of coagulation and complement factors correlated to WBC | Single time point (1 day)
  Individual composite mass spectrometric profile of 125 blood plasma factors containing the individual components of the coagulation system and the complement system correlated to leucocyte count (WBC)
Composite mass spectrometric profile of coagulation and complement factors correlated to maternal age | Single time point (1 day)
  Individual composite mass spectrometric profile of 125 blood plasma factors containing the individual components of the coagulation system and the complement system correlated to maternal age
Composite mass spectrometric profile of coagulation and complement factors correlated to placental weight | Single time point (1 day)
  Individual composite mass spectrometric profile of 125 blood plasma factors containing the individual components of the coagulation system and the complement system correlated to placental weight

CONTACTS AND LOCATIONS:
Overall Officials: Fabian B Fahlbusch, M.D., Principal Investigator — Department for Children- and Adolescent Medicine
Locations (1):
- Department of Pediatrics- and Adolescent Medicine, FAU Erlangen-Nuremberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No